CLINICAL TRIAL: NCT00373035
Title: Biomarkers of Prostate Cancer
Brief Title: Biomarkers in Patients Undergoing Transrectal Ultrasound Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU-85A03; CDR0000490117 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG03-628
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mass Spectrometry; Biopsy; High-Energy Shock Waves

INTERVENTIONS:
Genetic: proteomic profiling
Other: immunological diagnostic method
Other: laboratory biomarker analysis
Other: mass spectrometry
Procedure: biopsy
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Collecting and storing samples of blood and urine from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at biomarkers in patients undergoing transrectal ultrasound prostate biopsy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify unique proteins or peptides that are associated with prostate cancer by comparing the proteomic or metabolomic analysis of serum, plasma, and urine from patients with histological evidence of prostate cancer to those without prostate cancer (after transrectal ultrasound prostatic biopsy).

Secondary

* Collect seminal fluid from a subset of patients to test the hypothesis that the fluid collected from the "target organ of injury" in prostate cancer will have a higher signal of proteins/peptides that are different from those without cancer and may help guide the identification of these differences in the serum, plasma, and urine.

OUTLINE: This is a pilot study.

Patients undergo collection of serum, plasma, and urine for biomarker/laboratory analysis. Samples are examined by proteomic/metabolomic analysis (by mass spectrometry) and immunoassays. Patients then undergo a transrectal ultrasonography prostatic biopsy.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Indication for a transrectal ultrasonography prostatic biopsy (as part of normal patient care) due to elevated prostate-specific antigen, or abnormal digital rectal examination, or surveillance for prostate cancer

PATIENT CHARACTERISTICS:

* No prior or other concurrent malignancy except for curatively treated basal cell carcinoma of the skin
* No serious medical or psychiatric illness that would preclude informed consent
* No concurrent acute illness

PRIOR CONCURRENT THERAPY:

* No participation in another clinical trial within the past 30 days
* No more than one enrollment into this study

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Unique proteins or peptides associated with prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Torti, MD, MPH, Study Chair — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - SurroMed Incorporated, Menlo Park, California
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina